CLINICAL TRIAL: NCT02847299
Title: Comparison of a Hyperinflation Mode and Air Stacking on Neuromuscular Patients Under Volumetric Ventilation
Acronym: TWOTECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A00171-48
Record Dates: First submitted 2016-03-01; First posted 2016-07-28 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Neuromuscular Disease
Keywords: cough help; mechanical insufflation; mechanical ventilation; neuromuscular diseases; peak cough flow
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astral ventilator (Experimental): instrumental increase of cough peak flow with air stacking
  Interventions: Device: increase of cough peak flow ("Astral ventilator")
- Astral ventilator - mode kiné (Experimental): instrumental increase of cough peak flow with hyperinsufflation
  Interventions: Device: increase of cough peak flow ("Astral ventilator")

INTERVENTIONS:
Device: increase of cough peak flow ("Astral ventilator") — instrumental increase of cough peak flow with a ventilator by hyper-insufflation and with air stacking method

SUMMARY:
The purpose of the study is to compare the the efficacy and tolerance of 2 cough assistance techniques requiring no equipment other than the volumetric fan. The two methods are air-stacking and hyperinflation .

The study is a Cross-over, monocentric and open label study

DETAILED DESCRIPTION:
Primary outcome : Peak Expiratory Flow (PEF)

ELIGIBILITY:
Inclusion Criteria:

* age>18 years, neuromuscular disease,
* restrictive syndrome and/or cough peak flow < 270.l/mn and/or maximal expiratory pressure < 40 cm HO2,
* patient under non invasive ventilation
* steady state for at least one month
* written consent form given

Exclusion Criteria:

* bronchial congestion
* hemodynamic instability
* previous pneumothorax or emphysema bubbles
* Major bulbar dysfunction
* plan of legal protection
* pregnant or breastfeeding women
* no affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Peak cough flow | 1 year

SECONDARY OUTCOMES:
effective cough time | 1 year
inspired volume | 1 year
maximal expired volume | 1 year
respiratory comfort (Visual Analog Scale) | 1 year
subjective patient's effectiveness of cough (Visual Analog Scale) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frederic LOFASO, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Hopital R. Poincaré, Garches, Île-de-France Region, France

REFERENCES:
- [Background] Bach JR, Ishikawa Y, Kim H. Prevention of pulmonary morbidity for patients with Duchenne muscular dystrophy. Chest. 1997 Oct;112(4):1024-8. doi: 10.1378/chest.112.4.1024. PMID 9377912
- [Background] Tzeng AC, Bach JR. Prevention of pulmonary morbidity for patients with neuromuscular disease. Chest. 2000 Nov;118(5):1390-6. doi: 10.1378/chest.118.5.1390. PMID 11083691
- [Background] Gomez-Merino E, Bach JR. Duchenne muscular dystrophy: prolongation of life by noninvasive ventilation and mechanically assisted coughing. Am J Phys Med Rehabil. 2002 Jun;81(6):411-5. doi: 10.1097/00002060-200206000-00003. PMID 12023596
- [Background] Soudon P, Steens M, Toussaint M. A comparison of invasive versus noninvasive full-time mechanical ventilation in Duchenne muscular dystrophy. Chron Respir Dis. 2008;5(2):87-93. doi: 10.1177/1479972308088715. PMID 18539722
- [Background] Gomez-Merino E, Sancho J, Marin J, Servera E, Blasco ML, Belda FJ, Castro C, Bach JR. Mechanical insufflation-exsufflation: pressure, volume, and flow relationships and the adequacy of the manufacturer's guidelines. Am J Phys Med Rehabil. 2002 Aug;81(8):579-83. doi: 10.1097/00002060-200208000-00004. PMID 12172066
- [Background] Leger P, Paulus J. [Recommendations of HAS: Practical issues in home non-invasive ventilation in patients with neuromuscular disease]. Rev Mal Respir. 2006 Sep;23(4 Suppl):13S141-3. No abstract available. French. PMID 17057639
- [Background] Finder JD, Birnkrant D, Carl J, Farber HJ, Gozal D, Iannaccone ST, Kovesi T, Kravitz RM, Panitch H, Schramm C, Schroth M, Sharma G, Sievers L, Silvestri JM, Sterni L; American Thoracic Society. Respiratory care of the patient with Duchenne muscular dystrophy: ATS consensus statement. Am J Respir Crit Care Med. 2004 Aug 15;170(4):456-65. doi: 10.1164/rccm.200307-885ST. No abstract available. PMID 15302625
- [Background] Kang SW, Bach JR. Maximum insufflation capacity. Chest. 2000 Jul;118(1):61-5. doi: 10.1378/chest.118.1.61. PMID 10893360
- [Background] Bach JR. Update and perspective on noninvasive respiratory muscle aids. Part 2: The expiratory aids. Chest. 1994 May;105(5):1538-44. doi: 10.1378/chest.105.5.1538. No abstract available. PMID 8181348
- [Background] Boitano LJ. Management of airway clearance in neuromuscular disease. Respir Care. 2006 Aug;51(8):913-22; discussion 922-4. PMID 16867201
- [Background] Irwin RS, Boulet LP, Cloutier MM, Fuller R, Gold PM, Hoffstein V, Ing AJ, McCool FD, O'Byrne P, Poe RH, Prakash UB, Pratter MR, Rubin BK. Managing cough as a defense mechanism and as a symptom. A consensus panel report of the American College of Chest Physicians. Chest. 1998 Aug;114(2 Suppl Managing):133S-181S. doi: 10.1378/chest.114.2_supplement.133s. No abstract available. PMID 9725800
- [Background] Trebbia G, Lacombe M, Fermanian C, Falaize L, Lejaille M, Louis A, Devaux C, Raphael JC, Lofaso F. Cough determinants in patients with neuromuscular disease. Respir Physiol Neurobiol. 2005 Apr 15;146(2-3):291-300. doi: 10.1016/j.resp.2005.01.001. PMID 15766917
- [Background] Toussaint M, Boitano LJ, Gathot V, Steens M, Soudon P. Limits of effective cough-augmentation techniques in patients with neuromuscular disease. Respir Care. 2009 Mar;54(3):359-66. PMID 19245730
- [Background] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Background] Chatwin M, Ross E, Hart N, Nickol AH, Polkey MI, Simonds AK. Cough augmentation with mechanical insufflation/exsufflation in patients with neuromuscular weakness. Eur Respir J. 2003 Mar;21(3):502-8. doi: 10.1183/09031936.03.00048102. PMID 12662009
- [Background] Vianello A, Corrado A, Arcaro G, Gallan F, Ori C, Minuzzo M, Bevilacqua M. Mechanical insufflation-exsufflation improves outcomes for neuromuscular disease patients with respiratory tract infections. Am J Phys Med Rehabil. 2005 Feb;84(2):83-8; discussion 89-91. doi: 10.1097/01.phm.0000151941.97266.96. PMID 15668554
- [Background] Servera E, Sancho J, Zafra MJ, Catala A, Vergara P, Marin J. Alternatives to endotracheal intubation for patients with neuromuscular diseases. Am J Phys Med Rehabil. 2005 Nov;84(11):851-7. doi: 10.1097/01.phm.0000184097.17189.93. PMID 16244522
- [Background] Chatwin M, Simonds AK. The addition of mechanical insufflation/exsufflation shortens airway-clearance sessions in neuromuscular patients with chest infection. Respir Care. 2009 Nov;54(11):1473-9. PMID 19863831
- [Background] Bach JR. Mechanical insufflation-exsufflation. Comparison of peak expiratory flows with manually assisted and unassisted coughing techniques. Chest. 1993 Nov;104(5):1553-62. doi: 10.1378/chest.104.5.1553. PMID 8222823
- [Background] Lacombe M, Del Amo Castrillo L, Bore A, Chapeau D, Horvat E, Vaugier I, Lejaille M, Orlikowski D, Prigent H, Lofaso F. Comparison of three cough-augmentation techniques in neuromuscular patients: mechanical insufflation combined with manually assisted cough, insufflation-exsufflation alone and insufflation-exsufflation combined with manually assisted cough. Respiration. 2014;88(3):215-22. doi: 10.1159/000364911. Epub 2014 Aug 21. PMID 25171575
- [Background] Brito MF, Moreira GA, Pradella-Hallinan M, Tufik S. Air stacking and chest compression increase peak cough flow in patients with Duchenne muscular dystrophy. J Bras Pneumol. 2009 Oct;35(10):973-9. doi: 10.1590/s1806-37132009001000005. English, Portuguese. PMID 19918629
- [Background] Fauroux B, Guillemot N, Aubertin G, Nathan N, Labit A, Clement A, Lofaso F. Physiologic benefits of mechanical insufflation-exsufflation in children with neuromuscular diseases. Chest. 2008 Jan;133(1):161-8. doi: 10.1378/chest.07-1615. Epub 2007 Dec 10. PMID 18071020
- [Background] Kang SW, Kang YS, Sohn HS, Park JH, Moon JH. Respiratory muscle strength and cough capacity in patients with Duchenne muscular dystrophy. Yonsei Med J. 2006 Apr 30;47(2):184-90. doi: 10.3349/ymj.2006.47.2.184. PMID 16642546
- [Background] Sancho J, Servera E, Diaz J, Marin J. Efficacy of mechanical insufflation-exsufflation in medically stable patients with amyotrophic lateral sclerosis. Chest. 2004 Apr;125(4):1400-5. doi: 10.1378/chest.125.4.1400. PMID 15078752
- [Background] Winck JC, Goncalves MR, Lourenco C, Viana P, Almeida J, Bach JR. Effects of mechanical insufflation-exsufflation on respiratory parameters for patients with chronic airway secretion encumbrance. Chest. 2004 Sep;126(3):774-80. doi: 10.1378/chest.126.3.774. PMID 15364756